CLINICAL TRIAL: NCT05096351
Title: Immunological Reaction of the Recipient After Cold-stored Saphenous Venous Allograft (Bioprotec)
Acronym: REACIMALLOGV
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2021/EF-01
Record Dates: First submitted 2021-10-15; First posted 2021-10-27 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Allograft; Cold Temperature; Saphenous Vein
MeSH Terms: interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum, cell pellets, venous tissue
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with venous allograft
  Interventions: Other: Blood test

INTERVENTIONS:
Other: Blood test — Collection of blood samples at 1 and 6 months for HLA typing for donor and recipient antibodies

SUMMARY:
The study investigators propose to perform a blood test before and after allograft placement in all patients receiving a cold-stored venous allografts at the University Hospital of Nîmes to study the occurrence of FVFA-related ASD in these patients.

The aim of this work is to characterize a possible immune reaction generated by the implantation of venous allografts prepared according to the BIOPROTEC method. In case of a proven immune reaction, the study will allow a modification of our current attitude and to exclude patients potentially eligible for renal transplantation at the time of venous allograft placement, or to perform in these patients an allo-compatibility test with the venous allograft preoperatively and thus protect these patients from an increased risk of subsequent organ transplant rejection.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be a member or beneficiary of a health insurance plan
* Patients receiving a scheduled venous allograft within the CHU of Nîmes for an arterial bypass in the lower limb or an arteriovenous bypass in the upper limb within the framework of the creation of arteriovenous fistulas in dialysis patients, in the absence of available autologous venous material.

Exclusion Criteria:

* The subject is participating in a category 1 interventional study, or is in a period of exclusion determined by a previous study
* The subject has already been included in the study
* The subject refuses to participate
* It is impossible to give the subject informed information
* The patient is under safeguard of justice or state guardianship
* Patient previously having received a venous allograft or organ transplant
* Pregnant, parturient or breastfeeding patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving a scheduled venous allograft within the CHU of Nîmes for an arterial bypass in the lower limb or an arteriovenous bypass in the upper limb within the framework of the creation of arteriovenous fistulas in dialysis patients, in the absence of available autologous venous material.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-06-08 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Presence of donor specific antibodies after venous allograft | 1 month
  Presence/absence of donner anti-HLA antibodies in patient blood, detected using Luminex assay

SECONDARY OUTCOMES:
Allograft anomalies linked to allograft rejection | 1 month
  Inflammation, thrombosis, aneurysms progression
Allograft anomalies linked to allograft rejection | 6 month
  Inflammation, thrombosis, aneurysms progression

CONTACTS AND LOCATIONS:
Overall Officials: Elsa Faure, Principal Investigator — CHU Nimes
Locations (1):
- CHU de Nîmes, Nîmes, France